CLINICAL TRIAL: NCT04868279
Title: The Effect of Web-Based Interactive Nurse Support Program Based on Health Promotion Model on Healthy Living Behaviors and Self-Efficacy in Individuals Who Gain Weight After Bariatric Surgery: A Mixed Method Study
Brief Title: Weight Regain After Bariatric Surgery and Web-Based Interactive Nurse Support Program: Mixed Methods Research
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Ezgi Yildiz, Research Assistant, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SivasCumhuriyetU
Record Dates: First submitted 2021-04-23; First posted 2021-04-30 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Bariatric Surgery Candidate
Keywords: Weight regain after bariatric surgery; Health Promotion Model; Web-based interactive nurse support program; Healthy lifestyle behavior; Self-sufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In a randomized controlled study, blinding will be done in terms of statistician and reporting. Research data will be encoded and transferred to the computer without specifying the intervention and control group (for example; A group and B group). The analysis of these data coded in terms of groups will be done by a statistician. After the statistical analysis is done and the research report is written, the researcher will explain the coding for the intervention and control group. In this way, detection bias, statistical bias and reporting bias will be controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Gruop (Experimental): Web-based interactive nurse support program with the intervention group will continue for 3 months, the implementation will last 6 months in total. Individuals in the intervention group will be able to access the training content by accessing the website designated for the study from devices such as computers or mobile phones.
  Data collection forms will be applied to the intervention group 3 times in total, before starting the Web-based interactive nurse support program, at the end of the Web-based interactive nurse support program (in the 3rd month) and in the 6th month.
  Interventions: Behavioral: Web-Based Interactive Nurse Support Program Based on Health Promotion Model
- Control Group (No Intervention): Web-based interactive nurse support program will not be opened to the control group, only access to data collection tools will be provided.

INTERVENTIONS:
Behavioral: Web-Based Interactive Nurse Support Program Based on Health Promotion Model — Nursing education will be given on healthy behaviors such as nutrition, exercise, health responsibility and stress management according to the health promotion model. The researcher will make phone calls with the intervention group for 6 months (12 times in total), twice a month. During telephone interviews, individuals will be talking about the use of the website, the points that are not understood or need to be emphasized, their application of health promotion behaviors, the obstacles they experience during the application and the suggestions for this.
  Arms: Interventional Gruop

SUMMARY:
This study was planned to determine the effect of the web-based interactive nurse support program developed in line with the Health Promotion Model on healthy living behaviors and self-efficacy in individuals who gain weight after bariatric surgery. Mixed method is a research. The exploratory sequential design, one of the mixed research methods, will be used. The research will continue with the quantitative part starting with the qualitative part. The quantitative part of the research is a randomized controlled experimental study.

DETAILED DESCRIPTION:
This study was planned to determine the effect of the web-based interactive nurse support program developed in line with the Health Promotion Model on healthy living behaviors and self-efficacy in individuals who gain weight after bariatric surgery. Mixed method is a research. In the qualitative part of the study, factors that prevent individuals from developing health behaviors will be determined. In the quantitative part of the study, a web-based training program will be prepared in order to reduce the perception of disability in individuals towards health-enhancing behavior, to adopt a healthy behavior style and to increase their self-efficacy. The universe of the study will be individuals who had bariatric surgery in the general surgery service between 2015-2019 in a university hospital in Turkey and gained weight again. Qualitative interviews will be held face to face with the video method over the "Zoom" application. "Criterion sampling method", one of the purposeful sampling methods used in qualitative research, will be used. In the qualitative part of the research, the individual in-depth interview method will be selected, and the "Semi-Structured Interview Form" will be used as the data collection tool. Interviews with individuals will continue until data saturation is reached. All interviews will be recorded in digital format, transcribed and subsequently imported into the qualitative analysis software MAXQDA. The quantitative part of the research is a randomized controlled experimental study. Randomization will be done by a statistician other than the researcher. Power analysis was calculated using G * Power 3.1.9.7 program. With 80% effect size, 90% power and 0.05 significance level, the required sample size was determined as 28 individuals per group, and 56 individuals in total. It was decided to include 62 individuals, 31 individuals in the intervention group and 31 individuals in the control group, by taking 10% more of the calculated sample against the possibility of sample loss during the study. In the quantitative part of the study, the web-based interactive nurse support program will continue for 3 months, and the application will last for 6 months in total. A text message will be sent to their phones to remind individuals to use the website. The researcher will make phone calls with the intervention group for 6 months (12 times in total), twice a month. During telephone interviews, individuals will be talking about the use of the website, the points that are not understood or need to be emphasized, their application of health promotion behaviors, the obstacles they experience during the application and the suggestions for this. Healthy Lifestyle Behaviors Scale II, General Self-Efficacy Scale and Dutch Eating Behavior Questionnaire (DEBQ) will be used as measurement tools. Data collection forms will be applied to the intervention and control group three times in total, before starting the Web-based interactive nurse support program, at the end of the Web-based interactive nurse support program (in the 3rd month) and in the 6th month.After each assessment moment, the data obtained will be exported to the "Statistical Package for Social Sciences Software" (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* 18 years of age and above,
* at least two years past bariatric surgery and a history of weight gain,
* speaking Turkish,
* having no hearing, vision and understanding problems,
* independent in daily life activities,
* without dementia or alzheimer's diagnosis,
* literate individuals
* mobile phones and internet connections will be included in the study.

Exclusion Criteria:

* Individuals who are unable to use a computer or smart phone,
* have chronic illnesses,
* are pregnant,
* illiterate,
* who are currently participating in any healthy lifestyle program at least 2 months ago will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Healthy Lifestyle Behaviors Scale II | 6 months
  The scale measures health-promoting behaviors in relation to an individual's healthy lifestyle. The scale consists of 52 items in total. The scale has 6 sub-dimensions: health responsibility, physical activity, nutrition, spiritual development, interpersonal relationships, and stress management. For the whole scale, the lowest score is 52, the highest score is 208.
Dutch Eating Behavior Questionnaire (DEBQ) | 6 months
  The scale consists of 33 items. It has sub-dimensions such as emotional eating, restrictive eating, external eating. Items in the scale are evaluated with a 5-point Likert scale (1: never, 2: rarely, 3: sometimes, 4: often, 5: very often).
General Self-Efficacy Scale | 6 months
  It is a scale used to determine the general self-efficacy of adults. The scale, which consists of 17 items in total, is answered in the five-point Likert type. The score for each question ranges from 1 (none) to 5 (very good). The total score that can be obtained from the scale is between 17 and 85. The scale has 3 sub-dimensions in total. The increase in the total score of the scale indicates that the self-efficacy belief increases.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife KARAGÖZOĞLU, Prof. Dr, Study Director — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)